CLINICAL TRIAL: NCT01779869
Title: Development of a PET-MR Myocardial Perfusion Examination Using Regadenoson
Acronym: PET/MR-P
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Principal Investigator, Pamela Woodard, MD, Director of Center for Clinical Imaging Research (CCIR), Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PET/MR-Perfusion
Record Dates: First submitted 2013-01-23; First posted 2013-01-30 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-05

CONDITIONS: Ischemic Heart Disease
Keywords: PET MR myocardial perfusion imaging
MeSH Terms: conditions — Myocardial Ischemia | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group assignment - imaging (Experimental): All patients will undergo PET-MR myocardial perfusion imaging during rapid intravenous administration of 0.4 mg regadenoson.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Regadenoson 400 micrograms will be administered in a single IV bolus (<10 seconds) via an antecubital cannula and followed by 5 mL of saline flush. 10-20 seconds after the regadenoson is administered, 10 mCi of 13N-ammonia as a bolus, and 0.075 mmol/Kg of gadobenate dimeglumine MR contrast agent at a rate of 5 mL/sec followed by a 15 mL normal saline flush will be administered simultaneous, each into an antecubital vein, and a 15 min list-mode PET acquisition will be acquired simultaneously with the MR perfusion imaging.
  Other Names: Lexiscan

SUMMARY:
The objective for this pilot study is to develop an optimized, clinically usable myocardial PET-MR perfusion protocol and to determine which of all data potentially available should be acquired for a clinical myocardial perfusion examination. Hypothesis: The hypothesis is that high resolution, high sensitivity DCE MRI could replace the rest PET myocardial perfusion imaging, significantly decreasing examination time and patient radiation dose while maintaining the comprehensive reference-quality PET myocardial stress perfusion coverage.

The primary outcome will be comparison of diagnostic accuracy of each combination of imaging to detect clinically significant coronary artery stenosis (≥70% diameter stenosis).

DETAILED DESCRIPTION:
Simultaneous acquisition PET-MRI is a new technology that has the potential to significantly impact diagnostic patient care. It combines high signal resolution MRI anatomic imaging and PET biological measurements, with the added benefit of radiation dose reduction in comparison to PET-CT. As the incidence of false positive SPECT-MPI studies secondary to attenuation artifact is relatively high and MRI coverage of the left ventricular myocardium is limited, it is likely that one of the immediate applications of PET-MRI technology is myocardial ischemia assessment.

PET has long been considered the noninvasive reference standard for myocardial perfusion. However, delayed contrast enhanced (DCE) MRI is very sensitive for infarct detection. Indeed, both PET and MR imaging have the potential to provide comprehensive whole heart ischemia and infarct detection.

PET-MR technology, with its ability to obtain simultaneous perfusion information via both PET and MRI, has the potential to obtain multiple, possibly redundant, data sets. On the other hand, it also has the potential to combine the best of both techniques to provide a highly robust examination that is both shorter and of lower radiation dose than the standard myocardial PET perfusion examination. Optimization of a protocol is necessary to develop a comprehensive protocol without redundancy. Because of its single injection capability, regadenoson is ideally suited to a protocol that will assess and employ dual-modality myocardial perfusion data collection.

It is expected that the best candidates for PET-MR myocardial perfusion imaging will likely be a) patients whose body habitus suggests that their SPECT-MPI examination would be limited by attenuation artifact -- women with large breasts and patients (usually men) with abdominal obesity and/or b) patients who may have a smaller region of ischemia that might be missed on an MRI examinations with limited perfusion coverage.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had a clinically ordered rest/regadenoson single-isotope SPECT-MPI study within 10 days prior to cardiac PET-MRI examination
* Reversible perfusion abnormalities on SPECT imaging in at least 2 contiguous myocardial segments
* Patients for whom standard of care coronary ICA is planned

Exclusion Criteria:

* An clinical event (ie; worsening angina pectoris or myocardial infarction) occuring after the SPECT-MPI and before the cardiac MRI examination
* Myocardial revascularization occuring after the SPECT-MPI and before the cardiac MRI examination
* Contraindications to MR imaging (pacemaker, brain aneurysm clips, shrapnel, etc.)
* Renal insufficiency (GFR < 60 mL/min/1.73m2)
* Allergy or other contraindication to gadolinium-based MR contrast agent
* Second or third degree atrioventricular (AV) block
* Active asthma
* Seizures
* Current hypotension (<100/60)
* Current hypertension (>160/90)
* Pregnancy
* Breast feeding
* Use of caffeine, nicotine or over the counter cold medicines within 12 hours of the cardiac PET-MRI examination
* Use of the medication dipyridamole within 48 hrs of the cardiac PET-MRI examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela K Woodard, MD, BA, Principal Investigator — Washington University School of Medicine
Locations (1):
- Center for Clinical Imaging Research at Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
Analyzed data will be shared with other researchers after publication of manuscript.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Group Assignment - Imaging
Started | 16
Completed | 14
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: Individuals who had undergone a clinical SPECT stress test and were found to have ischemia in at least 2 continuous segments (based on a 17-segment model), and had been scheduled to undergo ICA for diagnostic and/or therapeutic considerations
Arm/Group | Single Group Assignment - Imaging
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Positive cardiac SPECT stress test (2 contiguous segments) [Count of Participants; unit: Participants] | 16
Scheduled to undergo ICA [Count of Participants; unit: Participants] | 16

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy of Cardiac PET/MRI Examination
Description: The accuracy of the cardiac PET and cardiac MR examination components of the PET/MRI, and the accuracy of the combined PET/MR examination, for ischemic heart disease will be compared to the accuracy of cardiac SPECT in patients who have had ICA as "truth" or the reference standard. To assess the accuracy of an abbreviated PET/MR examination, an additional accuracy analysis was made using only the stress PET perfusion imaging and the MR LGE data sets. The accuracy of this combined data set was also determined with ICA as "truth" or the reference standard. Accuracy is calculated as % difference = (experimental - true) x 100%.
Time Frame: PET/MRI imaging was performed within 10 days after SPECT-MPI examination
Population: Patients who completed the full PET-MR myocardial perfusion examination
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Single Group Assignment - Imaging
Number analyzed (Participants) | 16
percentage
  SPECT Accuracy | 50 [23 to 77]
  MR Accuracy | 64 [35 to 87]
  PET Accuracy | 61 [29 to 82]
  Combined PET/MR Accuracy | 64 [35 to 87]
  Abbreviated PET/MR | 64 [35 to 87]
Statistical Analysis 1: Comparison: Single Group Assignment - Imaging; Significance testing between the diagnostic accuracy of SPECT and PET, and SPECT and MR, and SPECT and PET/MR was performed by using chi square test. A P value < 0.05 was considered significant; Test type: Superiority — Accuracy was assessed compared to an imaging reference standard; p = 0.35, Chi-squared

ADVERSE EVENTS:
Time Frame: 24 hours after imaging
Arm/Group | Single Group Assignment - Imaging
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No